CLINICAL TRIAL: NCT05558553
Title: Are Neutrophil-Lymphocyte Ratio, Platelet-Lymphocyte Ratio, and Systemic Immune Inflammation Score Values Indicators for Postoperative Pain?
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Principal Investigator, Senay Canikli, medical specialist (Anesthesiology and Reanimation), Samsun University
Other Study IDs: 2022/4/11
Record Dates: First submitted 2022-09-24; First posted 2022-09-28 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Postoperative Pain Status of Patients Who Underwent Elective Laparoscopic Cholecystectomy
Keywords: Laparoscopic cholecystectomy; posoperative pain; neutrophil lymphocyte ratio; platelet lymphocyte ratio; systemic immune inflammation score; tramadol consumption

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postoperative pain status of patients who underwent elective laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Subject Researched:

Postoperative pain is a result of the inflammatory response to surgical trauma. Local inflammatory mediator response triggered by surgical incision, dissection, retraction, etc. causes an increase in nociceptor sensitivity and hyperalgesia, resulting in the perception of postoperative pain. With the acute phase response caused by surgical trauma, tissue damage is brought under control, infection is limited and the healing process begins. During the inflammatory response, the level of leukocytes in the blood also changes. Neutrophil/Lymphocyte ratio (NLR), Platelet/Lymphocyte ratio (PLR) and Systemic immune inflammation score (SII) are inexpensive and easily accessible biomarkers calculated from routine hemogram parameters and shown to be helpful in disease investigations and evaluation of treatment response. In this study, the relationship between biomarkers and postoperative pain status due to surgery will be investigated

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-75 years who underwent elective laparoscopic cholecystectomy.
2. Patients with ASA status1-2-3

Exclusion Criteria:

1. Emergency operated patients
2. Patients switched to open surgery
3. Patients allergic to tramadol
4. Those allergic to paracetamol
5. Those allergic to tenoxicam
6. Patients who cannot use the patient-controlled analgesia device
7. Those with hematological disorders
8. Those receiving immunosuppressive therapy
9. Those with inflammatory disease
10. Those with gastrointestinal tumors
11. Those with rheumatic disease
12. Those with uncontrolled diabetes
13. Those with chronic organ failure
14. Those who use corticosteroids
15. Opioid users
16. Those who have recently had an attack of cholecystitis, pancreatitis

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone elective laparoscopic cholecystectomy
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2022-09-18 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-24 (Actual)

PRIMARY OUTCOMES:
postoperative analgesic consumption | 24 hours

SECONDARY OUTCOMES:
postoperative pain score | 24 hours
  NRS 0-10 point

CONTACTS AND LOCATIONS:
Overall Officials: Şenay Canikli Adıgüzel, Study Director — responsibl investigator
Locations (2):
- Turkey (Türkiye) (2):
  - SAMSUN UNIVERSITY Samsun Training and research hospital, Samsun
  - Samsun Üniversity, Samsun

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be shared

REFERENCES:
- [Result] Tasargol O. A Prospective Study on the Predictability of Propofol Injection Pain. Cureus. 2020 Feb 10;12(2):e6945. doi: 10.7759/cureus.6945. PMID 32190496